CLINICAL TRIAL: NCT02308280
Title: A Phase II, Open-label Study of Bortezomib Following Nonmyeloablative Allogeneic Stem Cell Transplant in Patients With High-risk Multiple Myeloma
Brief Title: Nonmyeloablative Allogeneic Stem Cell Transplant Followed by Bortezomib in High-risk Multiple Myeloma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Dr Richard LeBlanc, Chair holder, Myeloma Canada Chair, Maisonneuve-Rosemont Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMR-MM-001
Record Dates: First submitted 2014-12-01; First posted 2014-12-04 (Estimated); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Multiple Myeloma; High-Risk Cancer
Keywords: High-risk myeloma; Non myeloablative allogeneic transplantation; Bortezomib
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib post-transplantation (Experimental): Non myeloablative allogeneic transplantation followed by Bortezomib for 1 year after a Bortezomib-based induction and autologous stem cell transplantation.
  Bortezomib: 1,3 mg/m2 subcutaneously every 2 weeks for 26 injections.
  Interventions: Drug: Bortezomib following nonmyeloablative allogeneic transplant

INTERVENTIONS:
Drug: Bortezomib following nonmyeloablative allogeneic transplant — Bortezomib 1,3 mg/m2 subcutaneously every 2 weeks for 1 year (26 injections) starting on day +120 from a non myeloablative sibling or 10/10 unrelated allogeneic transplantation
  Other Names: Velcade

SUMMARY:
Multiple myeloma is a morbid disease associated with a poor outcome, particularly those with high-risk cytogenetics. While standard therapies have modestly improved survival in these high-risk patients, myeloma remains incurable. To date, the only potential curative treatment remains allogeneic hematopoietic stem cell transplantation. However, the high incidences of toxicities including chronic GVHD and disease progression are currently the two most important obstacles to this therapy. Better approaches to maintain and improve benefits of allogeneic transplant, while decreasing toxicity, are urgently needed.

The investigators hypothesize that Bortezomib administration after non myeloablative allogeneic hematopoietic stem cell transplantation in high-risk myeloma patients might improved the outcome of these patients by decreasing myeloma relapse and the severity of chronic GVHD while preserving the graft-versus-myeloma effect. Our goal is to improve the poor clinical outcome of high-risk myeloma patients.

DETAILED DESCRIPTION:
To date, the only potential curative treatment for multiple myeloma remains allogeneic hematopoietic stem cell transplantation. Achievement of remission in myeloma patients allotransplanted with advanced disease, achievement of complete response in relapsed patients following infusion of donor leucocyte infusions, decreased incidence of relapse associated with chronic GVHD, better survival in myeloma patients who have relapsed after allogeneic transplant with rescue medication and production of an allo-immune response after allogeneic transplant, all support the existence of a graft-versus-myeloma effect. However, chronic GVHD participating to the morbidity and mortality of allogeneic transplantation, in addition to the significant relapse rate despite the transplantation are two important obstacles to this therapeutic modality in myeloma.

Bortezomib (VelcadeTM) is a dipeptidyl boronic acid-based reversible proteasome inhibitor. Several mechanisms of action have been proposed for its effects against multiple myeloma: direct induction of myeloma cells apoptosis, inhibition of NF-κB activation, reduction of myeloma cells adherence to the bone marrow microenvironment (decreasing drug resistance), inhibition of production, secretion and intracellular signalling of myeloma-mediators. It is one of the most effective drugs in the treatment of multiple myeloma. As consolidation treatment after autologous stem cell transplantation, the drug has been associated with an improvement in response rate and more importantly, in quality and depth of response. Maintenance treatment with Bortezomib after autologous transplantation has led to survival improvement, a benefit particularly obvious in myeloma patients with high-risk cytogenetics such as those carrying del(17p13).

In addition to its anti-myeloma properties, Bortezomib has immunomodulatory effects. Indeed, proteasome inhibitors affect several aspects of immune and inflammatory responses by interfering with antigen presenting cell function and effector cell function. Given its immunomodulatory properties, Bortezomib has recently been shown to be safe and effective in HLA-mismatched reduced-intensity conditioning transplantation as a GVHD prophylaxis.

This is a prospective phase II, open label, single institution study evaluating a novel treatment strategy in newly diagnosed multiple myeloma patients with high-risk disease or patients ≤ 50 years old. After an optimal Bortezomib-based induction treatment (VTD, CyBorD, RVD or PAD [in patients with plasma cell leukemia]) for a minimum of 4 cycles, followed by Melphalan ≥ 140 mg/m2 and autologous stem cell transplantation, eligible patients who accept to participate will be included in the study.

Within 6 months of autologous transplantation, patients will receive a non myeloablative allogeneic transplantation. Patients with a 6/6 compatible sibling donor will receive a conditioning regimen with Fludarabine 30 mg/m2 and Cyclophosphamide 300 mg/m2 per day for 5 days from day -8 to day -4 with 3 rest days before donor stem cell infusion on day 0. Patients without a sibling donor who have an 8/8 allele matched unrelated donor will receive a conditioning regimen of Fludarabine 30 mg/m2 per day for 3 days from day -4 to -2 and TBI 2 Gy on day -1 with donor stem cell infusion on day 0.

In sibling transplant recipients, GVHD prophylaxis will consist of Tacrolimus 3 mg p.o. BID starting on day -8, adjusted thrice weekly to obtain blood levels between 8-12 ng/mL. Tacrolimus tapering will start day +50 to be completed by day +100 in the absence of GVHD. In matched unrelated donor recipients, Tacrolimus will be initiated as in siblings, but started on day -4, and taper will be initiated on day +100 to be completed by day +180 in the absence of GVHD. MMF 15 mg/kg p.o. BID will be given from day +1 to +50 in sibling recipients. It will be given at same dose but TID from day +1 to +40, then tapered gradually until day +100 in matched unrelated donor recipients. Patients without progressive disease after allogeneic transplantation will receive Bortezomib 1.3 mg/m2 s.c. every 14 days ± 3 days starting on day +120, for a total of 26 doses (1 year treatment).

Patients will be followed regularly for disease evaluation, using the IMWG criteria. Toxicity will be evaluated using the NCI common terminology criteria for adverse events (CTCAE) version 4.0. Occurrence and severity of acute GVHD will be evaluated using the modified Glucksberg criteria. Chronic GVHD will be evaluated using the NIH criteria. The trial will be terminated when all patients have been followed for 5 years after allogeneic hematopoietic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years, inclusively
* Newly diagnosed multiple myeloma patients (according to IMWG criteria) with measurable disease at diagnosis, based on presence of any of the following:

  1. Serum intact immunoglobulin ≥ 10 g/L;
  2. Bence-Jones proteinuria ≥ 200 mg/day;
  3. Serum free light chain (sFLC) assay ≥ 100 mg/L (difference between involved and uninvolved FLC levels) and an abnormal sFLC ratio
* High-risk patients presenting any of the following:

  1. International Staging System (ISS) III;
  2. del(17p13), t(4;14) with ISS II or III, t(14;16), t(14;20) and chromosome 1 abnormalities by FISH. At this time, there is no international consensus on the threshold to consider these cytogenetic abnormalities as significant. For this study, investigators will consider arbitrarily a percentage ≥ 10% as significant.
  3. Plasma cell leukemia,defined as an absolute blood plasma cell count > 2 x 109/L and the presence of > 20% plasma cells among peripheral blood white cells;
  4. Patients ≤ 50 years, regardless of cytogenetics or ISS stage
* Having received a Bortezomib-containing regimen (VTD, CyBorD, VRD or PAD [in patients with PCL]) for a minimum of 4 cycles with ≥ PR.
* Received high-dose Melphalan ≥ 140 mg/m2 followed by autologous stem cell transplantation.
* Available HLA-identical sibling donor or 8/8 allele matched (HLA-A, -B, -C, -DR) matched unrelated donor

Exclusion Criteria:

* Failure to achieve at least PR with a Bortezomib-based induction therapy.
* Progressive disease at any time
* Having received tandem autologous stem cell transplantation.
* Having received maintenance or consolidation therapy with Bortezomib after ASCT. If delays to allogeneic transplant are expected, Lenalidomide at 10 mg die for a maximum of three months will be allowed after ASCT (initiated after day +90) and discontinued at least 14 days before the start of the conditioning regimen.
* Karnofsky score < 70% or comorbidity index HCT-CI > 3.
* Bilirubin > 2 x upper limit of normal (ULN) unless felt to be related to Gilbert's disease or hemolysis; AST and ALT > 2.5 x ULN; alkaline phosphatase > 5 x ULN.
* Peripheral neuropathy or neuropathic pain ≥ grade II.
* Poor organ function
* Known hypersensitivity to boron, mannitol or Bortezomib.
* Active infection with any of the following viruses: HIV, HTLV-1 or 2, hepatitis B (defined as HBsAg positivity) or hepatitis C (defined as anti-HCV positivity or HCV-RNA positivity).
* Presence of another malignancy with an expected survival estimated < 75% at 5 years (complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, complete resection of a ductal carcinoma in situ of the breast, presence of lobular carcinoma in situ of the breast, complete resection of carcinoma in situ of the cervix, or an in situ or low-risk prostate cancer after curative therapy are not exclusion criteria).
* Positive β-hCG pregnancy test. Female study participants who are surgically sterile (hysterectomy) or who have been postmenopausal for at least 12 consecutive months are automatically eligible for this criterion.
* Study participants not agreeing to remain abstinent or to practice double-barrier forms of birth control from trial screening through 90 days from the last dose of Bortezomib.
* Women who are lactating.
* Women of childbearing potential who are planning to become pregnant while enrolled in this study up to 30 days after the last Bortezomib injection.
* Participation in a trial with an investigational agent within 30 days prior to entry in the study.
* Inability to provide written informed consent prior to initiation of any study-related procedures, and inability, in the opinion of investigators, to comply with all requirements of the study
* Estimated probability to survive less than 6 months after allogeneic transplant.
* Suspicion of cardiac amyloidosis.
* Current history of drug and/or alcohol abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-09-27 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | At 2 years after allogeneic transplantation
  Progression-free survival is defined as the duration from start of the treatment to disease progression or death (regardless of cause of death), whichever comes first. A 2- sided confidence interval for this proportion will be computed. Minimal residual disease results from negativity to positivity using flow cytometry will not be used to define progression.

SECONDARY OUTCOMES:
Incidence of ≥ grade III non hematologic toxicity (including ≥ grade II peripheral neuropathy) and incidence of ≥ grade IV hematologic toxicity | At each medical visit up to 5 years from allogeneic transplantation
  Non hematologic toxicity and hematologic toxicity will be graded according to CTCAE v.4.0.
Cumulative incidence of grade I-IV and grade II-IV acute GVHD | At day 100 days, 6 months and 1 year after allogeneic transplantation
  Acute GVHD will be graded according to modified Glucksberg criteria
Cumulative incidences of chronic GVHD | At 1 and 2 years after allogeneic transplantation
  Chronic GVHD will be evaluated according to NIH criteria
Maximum grades of acute and chronic GVHD | At each medical visit up to 5 years from allogeneic transplantation
  Acute and chronic GVHD evaluation will based on modified Glucksberg and NIH criteria, respectively
Response rates and quality of responses | Before allogeneic transplantation, before bortezomib, 1 year after bortezomib, then every 8 to 12 weeks up to 5 years from allogeneic transplantation
  Response categories will be assessed based on the IMWG criteria
Nonrelapse mortality | At 100 days and 2 years
  Nonrelapse mortality is defined as time to deaths without relapse or recurrence. Deaths from any cause without prior progression are events.
Overall survival | At 2 years
  Overall survival is defined as time to death, irrespective of the cause.
Incidence of relapse | At 2 years
  Relapse is defined as progression of the disease previously treated, based on the IMWG criteria.
Minimal residual disease on bone marrow using multiparametric flow cytometry | Before the allogeneic transplantation, before Bortezomib administration (day +120), at 3, 6, 9, 12, 15, 18, 21 and 24 months from day +120 of the allogeneic transplantation
  From ≥ 5 million events, specimens with less than 50 aberrant phenotype plasma cells will be considered as MRD negative
Quality of life after allogeneic transplantation | Evaluated before allogeneic transplantation, at 100 days from transplantation, before Bortezomib administration, then every 3 months up to 5 years from allogeneic transplantation
  Quality of life will be assessed prospectively by the EORTC QLQ-MY20, EORTC QLQ-C30 (version 3) and FACT-BMT (version 4) questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Richard LeBlanc, M.D., Principal Investigator — Hôpital Maisonneuve-Rosemont, affiliated to University of Montreal
Locations (1):
- Hôpital Maisonneuve-Rosemont, Montreal, Quebec, Canada